CLINICAL TRIAL: NCT07320781
Title: Role of Preoperative Tapentadol in Reduction of Perioperative Analgesic Requirement After Breast Conservative Surgery in Cancer Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-23-20
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Tapentadol; Breast Cancer Surgery; Morphine
MeSH Terms: conditions — Breast Neoplasms | interventions — Tapentadol

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Care Provider
Masking Description: The patient and doctor providing anesthesia were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tapentadol (Active Comparator): Control drug (Tapentadol )
  Interventions: Drug: Tapentadol
- Placebo (Placebo Comparator): Placebo sodium bicarbonate/ peppermint oil tablet
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tapentadol — 75 mg oral tapentadol given 1 hour before surgery in control group and placebo tablet was given in Group B. Intraoperative and post operative morphine consumption and pain scores at 1,2,3,4 hours were calculated.
  Arms: Tapentadol
Other: Placebo — Placebo tablet was given in group B.
  Arms: Placebo

SUMMARY:
This study evaluated the preemptive analgesic efficacy of Tapentadol in reducing peri operative analgesic requirements among patients undergoing breast cancer surgery.

DETAILED DESCRIPTION:
A double blinded prospective RCT was conducted with 70 patients undergoing breast cancer surgery with 35 patients being studied with Administrated drug & other 35 as placebo. Intraoperative & postoperative morphine consumption was calculated and documented.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years
2. ASA 1,2,3
3. Patients scheduled for breast conservation surgery -

Exclusion Criteria:

1. Patient refusal
2. CKD greater than 3
3. BMI greater than 35
4. Known drug allergy -

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females.
Enrollment: 70 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Intraoperative and postoperative morphine consumption | During the course of surgery and up to 4 hours surgery
  During the course of surgery and up to 4 hours surgery Intraoperative and postoperative morphine consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Allah Ditta Ashfaq, Study Director — Shaukat Khanam Memorial Cancer Hospital & Research Centre LAHORE
Locations (1):
- SKMCH & RC Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD. Due to confidentiality of patients data.